CLINICAL TRIAL: NCT06309290
Title: Prehabilitation Based on Resistance-exercise Training in Women With Breast Cancer Undergoing Neoadjuvant Therapy: From Molecular Mechanism to Clinical Benefits
Brief Title: Prehabilitation With Resistance-exercise Training for Breast Cancer Neoadjuvant Therapy
Acronym: NEO STRONG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de La Frontera (Other)
Responsible Party: Principal Investigator, Gabriel Nasri Marzuca-Nassr, Principal Investigator, Universidad de La Frontera
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FAPESP-UFRO
Record Dates: First submitted 2024-02-29; First posted 2024-03-13 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Prehabilitation; Breast Cancer; Postmenopause; Resistance Training
Keywords: Prehabilitation; Breast neoplasm; Strength Training; Skeletal muscle; Muscle strength
MeSH Terms: conditions — Breast Neoplasms | interventions — Preoperative Exercise; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prehabilitation intervention program (Experimental): All volunteers be subjected to 16 - 20 weeks of full body resistance exercise training (2 times per week. However, usual care program.
  Interventions: Other: Prehabilitation with resistance-exercise training
- Usual Care Program (Active Comparator): All volunteers be subjected usual care (diagnosis confirmation, chemotherapy treatment planning and an initial education session).
  Interventions: Other: Usual care program

INTERVENTIONS:
Other: Prehabilitation with resistance-exercise training — The volunteers in the intervention group will be subjected to 16 - 20 weeks of whole-body resistance-type exercise training (2x/wk).
  Other Names: Prolonged resistance-type exercise training; Prehabilitation
  Arms: Prehabilitation intervention program
Other: Usual care program — The volunteers in the intervention group will be subjected to usual care (diagnosis confirmation, chemotherapy treatment planning and an initial education session).
  Other Names: Standard therapy
  Arms: Usual Care Program

SUMMARY:
Breast cancer stands as the foremost cause of cancer-related deaths among women worldwide, with the highest incidence of any cancer type. The choice of therapeutic interventions hinges upon factors like cancer stage, cell subtype, and tumor size. Consequently, individuals with more aggressive tumors, such as HER+2 and Triple Negative, or larger tumors often undergo neoadjuvant chemotherapy before breast surgery. However, these anticancer treatments come with side effects like cancer-related fatigue, reduced functional capacity, and changes in body composition, notably skeletal muscle atrophy. Skeletal muscle loss correlates with heightened mortality rates, cardiotoxicity, and diminished quality of life, underscoring the need for early therapeutic interventions. One such promising strategy is prehabilitation, which involves resistance-exercise training aimed at bolstering skeletal muscle mass from the outset of the disease, even preceding breast surgery. Resistance-exercise training has shown favorable effects on women undergoing adjuvant therapy or survivors of breast cancer, however, its molecular and clinical effects in women with breast cancer undergoing neoadjuvant therapy are unknown.

DETAILED DESCRIPTION:
Hypothesis: Prehabilitation based on resistance-exercise training before surgery in women with breast cancer undergoing neoadjuvant therapy increases skeletal muscle mass compared with usual care.

Secondary, prehabilitation based on resistance-exercise training before surgery in women with breast cancer undergoing neoadjuvant therapy generates better results in body composition, physical performance, clinical parameters (serious adverse events, hospital readmission, infection, complications), physiological parameters and quality of life at one-month hospital discharge compared to usual care.

Objective: To determine the effects of prehabilitation based on resistance-exercise training versus usual care, before and after breast surgery, on skeletal muscle mass in women with breast cancer undergoing neoadjuvant chemotherapy.

Methodology: A single-blind, randomized controlled clinical trial will be developed. Sixty-eight postmenopausal women with stage I, II and III breast cancer with HER2+ type breast tumor and Triple negative breast cancer undergoing neoadjuvant therapy and with an indication for breast surgery will be divided into two groups: usual care (CONTROL, n=34) versus Prehabilitation (P-REHAB, n=34). All participants will receive an education session 20 weeks before surgery + neoadjuvant chemotherapy for 16-20 weeks as is normally done for this type of patien. Only participants in the P-REHAB group will undergo 16-20 weeks of whole-body resistance-exercise training (twice a week). At baseline, after prehabilitation program and 4 weeks after surgery, the cross-sectional area of the quadriceps muscle and of the muscle region at lumbar level 3 will be determined by CT-Scan. Also, fasting blood samples will be obtained to measure biochemical and molecular markers (e.g. miRNAs). Maximal strength will be determined by 1 repetition maximum (1RM) leg press, leg extension, lat pull down, chest press, horizontal row, and handgrip. In addition, physical performance will be assessed with the short physical performance battery (SPPB), functional capacity with the 6-minute walk test, quality of life with the BR23 questionnaire, and cancer-related fatigue with the Brief Fatigue Inventory scale at the same time points. Finally, samples from tumor breast cancer and pectoralis muscle will be obtained on the day of breast surgery.

Expected results: It is expected that prehabilitation based on resistance-exercise training results in increased muscle mass in women with breast cancer undergoing neoadjuvant chemotherapy compared to participants receiving usual care. Also, it is expected that this intervention before surgery in women with breast cancer undergoing neoadjuvant therapy will generate better results in clinical parameters (serious adverse events, hospital readmission, infection, complications) and quality of life one month after hospital discharge compared to usual care . These results will allow the creation of local, regional, national and international strategies to combat the adverse effects of breast cancer and its antineoplastic treatment, especially in women with more aggressive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with breast cancer in stages I, II and III with luminal breast tumor, HER2+ or TNBC
* Indication for neoadjuvant chemotherapy
* Candidates for curative breast surgery
* Body mass index: 18.5 <BMI <30 kg/m2
* Sedentary (does not perform scheduled or planned physical activity ≥ 2 times a week)
* Willingness to participate in the study and follow the proposed prehabilitation scheme.

Exclusion Criteria:

* Present comorbidities that interact with the metabolism and mobility of the muscles of the body and that do not allow the (safe) performance of strength exercises (e.g., debilitating arthritis, all neurological disorders, paralysis, among others).
* Severe or uncontrolled cardiovascular disease, cardiac ejection fraction less than 50%
* Previous antineoplastic treatment
* Use of nutritional supplements (leucine, glutamine, casein, whey protein, fatty acids and creatine).

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 68 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in skeletal muscle mass (measured via Computed tomography (CT) scan) | Before training (week 0), and after training (up to 20 weeks) and 4 weeks post surgery
  Cross-sectional area of the quadriceps via single-slice CT scan

SECONDARY OUTCOMES:
Change in arms and legs strength (measured via 1-Repetition Maximum (1RM) testing) | Before training (week 0), and after training (up to 20 weeks) and 4 weeks post surgery
  Maximal strength assessment via 1RM testing of horizontal row, lat pull down, chest press, leg press, and leg extension)
Change in hand grip strength (measured via JAMAR handheld dynamometer) | Before training (week 0), and after training (up to 20 weeks) and 4 weeks post surgery
  Maximal strength assessment via 1RM testing of JAMAR handheld dynamometer.
Change in physical performance measured via Short physical performance battery | Before training (week 0), and after training (up to 20 weeks) and 4 weeks post surgery
  Measurement of physical performance via SPPB Short physical performance battery (0 to 12 points, whether higher scores mean a better outcome).
Change in points quality of life measured via questionnaire European Organisation for Research and Treatment of Cancer (EORTC QLQ-C30) | Before training (week 0), and after training (up to 20 weeks) and 4 weeks post surgery
  Measurement of quality of life via EORTC QLQ-30, this questionnaire has 30 question covering functional state and cancer related symptoms. Besides, there are two specific question covering the "overall health" and "overall quality of life". The scores obtained are standardized and a score between 0 and 100 is obtained. High values on the global health and functional status scales indicate a better quality of life. However, high values on the symptom scale indicate a lower quality of life
Change in points Brief fatigue inventory (BFI) | Before training (week 0), and after training (up to 20 weeks) and 4 weeks post surgery
  The instrument consists of nine items, each rated on a scale from 0 to 10, aimed at assessing fatigue. By averaging the scores of all items, a fatigue score is derived, wherein higher values signify more severe fatigue.
Change in microgram per milliliter (µg/ml) of Human Insulin via ELISA | Before training (week 0), and after training (up to 20 weeks) and 4 weeks post surgery
  Measurement in blood samples, the insulin will evaluate by ELISA using the Human Insulin ELISA Kit, following the manufacturer's recommendations
Change in pathological complete response rate | Before training (week 0), and after training (up to 20 weeks)
  Measured according to Sataloff criteria.
Change quantification proteins | Before training (week 0), and after training (up to 20 weeks)
  It will be measured from a muscle sample obtained at the time of surgery using the western blot technique.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel N Marzuca-Nassr, PT, MSc, PhD, Principal Investigator — Universidad de La Frontera
Locations (2):
- Chile (2):
  - Fundación Arturo López Pérez, Santiago
  - Department of Rehabilitation Sciences, Faculty of Medicine, Universidad de La Frontera. Temuco, Chile, Temuco

IPD SHARING:
Plan to Share IPD: No